CLINICAL TRIAL: NCT01549574
Title: A Phase 1, Open Label, Single Dose, Randomized, Cross-Over Study To Estimate The Effect Of Esomeprazole On The Pharmacokinetics Of Crizotinib In Healthy Volunteers
Brief Title: Drug Drug Interaction Study Of Crizotinib With Esomeprazole.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A8081035
Record Dates: First submitted 2012-02-25; First posted 2012-03-09 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: crizotinib; pharmacokinetics; esomeprazole; proton pump inhibitor; drug drug interaction; healthy volunteers
MeSH Terms: interventions — Crizotinib; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- crizotinib/crizotinib+esomeprazole crossover (Experimental): Each subject in this study will receive two treatments (A and B) separated by at least 14 days of washout period. Treatment A is a 250 mg single oral dose of crizotinib administered in a fasted state as 1x 250 mg Formulated Capsule. Treatment B consists of 40 mg daily esomeprazole dose from Day 1 to Day 5 and a 250 mg single oral dose of crizotinib administered in a fasted state as 1x 250 mg Formulated Capsule on Day 5.
  Interventions: Drug: crizotinib; Drug: esomeprazole

INTERVENTIONS:
Drug: crizotinib — Each subject in Treatment A will receive a 250 mg single oral dose of crizotinib administered in a fasted state as 1x 250 mg Formulated Capsule on Day 1 and each subject in Treatment B will receive a 250 mg single oral dose of crizotinib administered in a fasted state as 1x 250 mg Formulated Capsule on Day 5
Drug: esomeprazole — Each subject in Treatment B will receive 40 mg daily dose of esomeprazole from Day 1 to Day 5

SUMMARY:
This is an open-label, randomized, cross-over, single dose study in healthy volunteers to evaluate the potential effect of esomeprazole, a proton pump inhibitor, on the pharmacokinetics of crizotinib. Each subject enrolled will receive two single oral doses of crioztinib with or without esomeprazole separated by a washout period of at least 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female of non childbearing potential subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG or clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of Screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half lives preceding the first dose of study medication.
* Screening supine blood pressure >= 140 mm Hg (systolic) or >=90 mm Hg (diastolic), on a single measurement (confirmed by a single repeat, if necessary) following at least 5 minutes of rest.
* Screening 12 lead ECG demonstrating QTc >450 or a QRS interval >120 msec at Screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.
* Pregnant or nursing females; females of childbearing potential, including those with tubal ligation.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication. Herbal supplements and hormone replacement therapy must be discontinued 28 days prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of =< 1 g/day. Limited use of non prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* A positive serology for Hepatitis B or Hepatitis C.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Plasma AUCinf [area under the plasma concentration-time profile from time 0 to infinite time] for crizotinib | 2 months
Plasma Cmax [maximum observed concentration] for crizotinib | 2 months

SECONDARY OUTCOMES:
Plasma AUClast [area under the plasma concentration-time profile from time zero to the time of the last quantifiable concentration] for crizotinib | 2 months
Plasma Tmax [time for maximum observed concentration] for crizotinib | 2 months
Plasma t1/2 [terminal half-life] for crizotinib | 2 months
Plasma CL/F [apparent oral clearance] for crizotinib | 2 months
Plasma Vz/F [apparent volume of distribution] for crizotinib | 2 months
Plasma AUClast for metabolite (PF-06260182) if appropriate | 2 months
crizotinib/metabolite AUClast ratio if appropriate | 2 months
Plasma AUCinf for metabolite (PF-06260182) if appropriate | 2 months
crizotinib/metabolite AUCinf ratio if appropriate | 2 months
Plasma Cmax for metabolite (PF-06260182) if appropriate | 2 months
crizotinib/metabolite Cmax ratio if appropriate | 2 months
Plasma Tmax for metabolite (PF-06260182) if appropriate | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- [Derived] Xu H, O'Gorman M, Matschke K, Boutros T, Brega N, Tan W, Bello A. Evaluation of Proton Pump Inhibitor Esomeprazole on Crizotinib Pharmacokinetics in Healthy Participants. Clin Pharmacol Drug Dev. 2022 Jan;11(1):34-42. doi: 10.1002/cpdd.1032. Epub 2021 Nov 26. PMID 34825782
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081035&StudyName=Drug%20Drug%20Interaction%20Study%20Of%20Crizotinib%20With%20Esomeprazole.